CLINICAL TRIAL: NCT00645242
Title: An Open Label, Multicenter Trial Of Diflucan (Fluconazole) For 6 Weeks Given Once Daily To Pediatric Patients With Tinea Capitis
Brief Title: A Study Of Diflucan In Children With Ringworm Of The Scalp
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0561017
Record Dates: First submitted 2008-03-25; First posted 2008-03-27 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Tinea Capitis
MeSH Terms: conditions — Tinea Capitis | interventions — Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental)
  Interventions: Drug: fluconazole

INTERVENTIONS:
Drug: fluconazole — Fluconazole oral suspension 6 mg/kg/day for 6 weeks followed by 4 weeks without treatment

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of fluconazole for the treatment of tinea capitis in pediatric patients aged 3 to 12 years.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (aged 3-12 years)
* Clinical diagnosis of tinea capitis
* Direct microscopy (KOH) positive for fungal elements within or outside hair shaft

Exclusion Criteria:

* Negative baseline KOH
* Liver disease

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 185 (Estimated)
Dates: Start 2002-11; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Combined clinical and mycological outcome at Week 6 | Week 6

SECONDARY OUTCOMES:
Clinical outcome based on signs and symptoms at Weeks 3, 6, and 10 | Weeks 3, 6, and 10
Combined clinical and mycological outcome at Weeks 3 and 10 | Weeks 3 and 10
Mycological outcome based on culture results at Weeks 3, 6, and 10 | Weeks 3, 6, and 10
Culture results at Weeks 3, 6, and 10 | Weeks 3, 6, and 10

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- United States (25):
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Martinez, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Evanston, Illinois
  - Pfizer Investigational Site, Gretna, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Fridley, Minnesota
  - Pfizer Investigational Site, Bridgeton, Missouri
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Garner, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Murfreesboro, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Norfolk, Virginia
- Puerto Rico (2):
  - Pfizer Investigational Site, Carolina
  - Pfizer Investigational Site, Ponce

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0561017&StudyName=A%20Study%20Of%20Diflucan%20In%20Children%20With%20Ringworm%20Of%20The%20Scalp